CLINICAL TRIAL: NCT02831426
Title: Prospective Multicentric Randomized Comparison of an Acellular Dermal Matrix Versus a Synthetic Mesh in Pre-pectoral Implant Based Breast Reconstruction
Brief Title: Pre-pectoral Breast Reconstruction PART 2
Acronym: PreBRec
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Kovacs, PhD, FRCS, Guy's and St Thomas' NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCTBU022016
Record Dates: First submitted 2016-06-29; First posted 2016-07-13 (Estimated); Last update posted 2016-10-03 (Estimated); Status verified 2016-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tissue Expansion Devices

ARMS (2):
- ADM two-stage reconstruction (Active Comparator): Two-stage with Acellular Dermal Matrix (CELLIS® Breast). Tissue Expander A, Pre-pectoral, subcutaneous, two-stage reconstruction by means of TE supported by ADM
  Interventions: Device: Two-stage with Acellular Dermal Matrix (CELLIS® Breast)
- TCPM two-stage reconstruction (Experimental): Two-stage with Titanium Coated Polypropylene Mesh (TiLOOOP® Bra). Tissue Expander B, Pre-pectoral, subcutaneous, two-stage reconstruction by means of TE supported by TCPM
  Interventions: Device: Two-stage with Titanium Coated Polypropylene Mesh (TiLOOOP® Bra)

INTERVENTIONS:
Device: Two-stage with Acellular Dermal Matrix (CELLIS® Breast) — After mastectomy, an immediate reconstruction will be performed by means of a tissue expander, of any shape and type available, positioned in a subcutaneous, pre-pectoral, position. The tissue expander will be held in place by an ADM (CELLIS® Breast, MECCELLIS BIOTECH, 40 rue Chef de Baie, 17000, La Rochelle FRANCE) either completely wrapped around it or just covering its anterior surface. After at least 6 months a TE/implant exchange procedure will be performed with a synchronous fat grafting procedure to ameliorate the skin flap thickness and softness over the medial border and upper pole. Fat grafting will be performed with the wash and filter principle technique of handling the harvested fat tissue.
  Other Names: Tissue Expander two-stage reconstruction with ADM; Tissue Expander / Implant exchange; Fat grafting
  Arms: ADM two-stage reconstruction
Device: Two-stage with Titanium Coated Polypropylene Mesh (TiLOOOP® Bra) — After mastectomy, an immediate reconstruction will be performed by means of a tissue expander, of any shape and type available, positioned in a subcutaneous, pre-pectoral, position. The tissue expander will be held in place by a Titanium Coated Polypropylene Mesh (TiLOOOP® Bra, pfm medical, ag Wankelstraße 60 ,50996 Köln GERMANY) either completely wrapped around it or just covering its anterior surface. After at least 6 months a TE/implant exchange procedure will be performed with a synchronous fat grafting procedure to ameliorate the skin flap thickness and softness over the medial border and upper pole. Fat grafting will be performed with the wash and filter principle technique of handling the harvested fat tissue.
  Other Names: Tissue Expander two-stage reconstruction with TCPM; Tissue Expander / Implant exchange; Fat grafting
  Arms: TCPM two-stage reconstruction

SUMMARY:
The rationale for present trial conception and design moves forward from the assumption that a subcutaneous, pre-pectoral reconstruction by means of soft tissue replacement devices is feasible, safe and giving rewarding results when compared to the standard retro-pectoral technique. Ahead of that, the trial aims to test if there is a difference in the outcomes between a biological and a synthetic material when placed as a support under the mastectomy skin flaps, both in terms of immediate complications and of long-term results.

DETAILED DESCRIPTION:
This phase III randomized clinical trial will be investigating the Two-stage, using Tissue Expander (TE) pre-pectoral reconstructions.

The trial will comprise two arms:

PRE-PECTORAL technique with a biological Acellular Dermal Matrix (ADM) prosthesis coverage and support + FAT GRAFTING VS PRE-PECTORAL technique with a synthetic Titanium Coated Polypropylene Mesh (TCPM) prosthesis coverage and support + FAT GRAFTING

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will entail cases of conservative mastectomies (skin-sparing mastectomy SSM, nipple-sparing mastectomy NSM and skin-reducing mastectomy SRM), both prophylactic and therapeutic.

Included patients baseline characteristics will be:

* age 18-80 years old
* BMI between 18.5 and 35.
* Former smokers (up until 3 weeks before surgery)
* hypertension at oral medications
* diabetes
* previous breast surgery
* previous breast and chest wall radiation therapy will be allowed.

Exclusion Criteria:

* T4 and metastatic breast cancers
* obese patients (BMI over 35)
* currently smoking patients (within 3 weeks before surgery)
* refusal to sign the consent
* severe comorbidities requiring a chronic therapy (renal failure, heart failure, cardiovascular diseases, pulmonary diseases, hepatic diseases, and metabolic diseases).

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Rate in percentage of surgical complications | up to 6 months
  Surgical outcomes will be evaluated considering the rate in percentage of cases affected by the following complications among total number:
  surgical site infection (any infection requiring an antibiotic therapy, either oral or intravenous), wound dehiscence, seroma (any fluid collection requiring aspiration for more than a month from mastectomy), nipple/skin necrosis (either partial or complete), hematoma, red breast syndrome, with their reintervention rate. Rates will be compared between the two groups
Rate in percentage of technique failure | up to 6 months
  The failure rate, as percentage, will be compared between the two arms:
  failure will be the prosthesis (implant or TE) loss rate (reintervention with prosthesis removal) among overall number of prostheses implanted.

SECONDARY OUTCOMES:
Objective quality of life assessment with Baker scale for capsular contracture | at 2 years from mastectomy
  Long-term outcomes, after two years from mastectomy and at least 3 months from TE/implant exchange, in quality of life will entail first of all an objective assessment: such evaluation will include the capsular contracture rate, with the assessment of the reintervention rate for amelioration or for a reconstructive strategy change. Among these objective evaluations, any possible short-term complications after second-stage procedure will be investigated.
Objective quality of life assessment with cosmetic evaluation on pictures with a Likert scale for scoring | at 2 years from mastectomy
  A third party objective evaluation will be carried out by a group of a surgeon, a nurse and a lay person from a different center from that one where every single case was performed. This third party evaluation will assess the cosmetic outcome based on medical photographic files, giving a score for each patient. Scores from the two arms will be compared.
Subjective quality of life assessment with BREAST-Q questionnaire (Memorial Sloan-Kettering Cancer Center and The University of British Columbia © 2006, all rights reserved) | at 2 years from mastectomy
  After 2 years from mastectomy and at least 3 months from TE/implant exchange a subjective evaluation will be carried out with BREAST-Q score (scores from the two arms will be transformed in 100 scale, summed and compared as median)

OTHER OUTCOMES:
Cost-efficiency analysis with comparison of cost in money of the two arms | at 3 years from mastectomy
  Analysis of costs with comparison of the two arms will be carried out considering all costs from procedures and materials to possible late reinterventions to resolve complications and problems
Rate in percentage of complications in the sub-group of irradiated patients | at 3 years from mastectomy
  An analysis of a specific subgroup of patients will be carried out, namely those previously submitted to a breast irradiation and those submitted to a post-mastectomy radiation therapy. Analysis of short-terms failures and long-term problems with change in reconstruction strategy will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Breast Surgery Unit, Guy's and St Thomas' Hospital NHS Trust, London, United Kingdom